CLINICAL TRIAL: NCT07219758
Title: RECANA OUS - Recana Thrombectomy Catheter System for Venous Obstruction and Occlusion Study (RECANA-OUS-UK)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intervene, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN014
Record Dates: First submitted 2025-10-17; First posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Venous Obstruction
Keywords: chronic venous disease; chronic venous insufficiency; CEAP classification of C3 or greater; flow-limiting venous outflow obstruction; post-thrombotic syndrome (PTS); venous inflow/outflow obstruction
MeSH Terms: conditions — Postthrombotic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Open-label (Experimental): prospective, non-randomized treatment with the Recana Thrombectomy Catheter System
  Interventions: Device: Recana Thrombectomy Catheter System

INTERVENTIONS:
Device: Recana Thrombectomy Catheter System — recanalization and debulking of obstructions and occlusions within stented and non-stented segments in veins

SUMMARY:
The goal of this clinical investigation is to learn if the Recana Thrombectomy Catheter System can treat chronic venous obstruction and occlusion in participants with symptomatic post-thrombotic venous inflow/outflow obstruction. The main questions the clinical investigation aims to answer are:

1. primary safety endpoint: procedural events defined as the rates of all adverse events occurring up to 30 days post-index procedure
2. primary efficacy endpoint: percent (%) lumen gain during the index procedure, which is measured using intravascular ultrasound (IVUS) at the time of the procedure (perioperative/periprocedural)

Participants are screened and qualified for the clinical investigation. Qualifed participants (those that meet all eligibility criteria) will undergo treatment with the Recana Thrombectomy Catheter System. Participants are assessed at the following timepoints: 30, 90, 180 and 365 days post-procedure.

DETAILED DESCRIPTION:
STUDY DESIGN: The RECANA Study is a prospective, non-randomized, safety and performance (efficacy) study to evaluate participants treated with the Recana Thrombectomy Catheter System for the treatment of symptomatic post-thrombotic venous inflow/outflow obstruction.

STUDY OVERVIEW: Potential participants who pass pre-screening and are willing to participate in the study will be asked to sign the study Informed Consent Form before any study-specific tests or procedures are performed or for any study specific evaluations not considered standard of care that need to be performed to assess eligibility.

Eligible participants may undergo the index procedure. Adverse events are assessed starting on the day of the index procedure (considered Time 0) through 365 days post-procedure. All participants enrolled in the study are evaluated at screening/baseline, index procedure through hospital discharge, 30-days, 90-days,180 days and 365 days post-procedure. Duplex ultrasound, clinical assessments, quality of life, adverse events and concomitant medications are assessed at each follow-up visit.

STUDY POPULATION: Patients with symptomatic post-thrombotic venous inflow/outflow obstruction.

STUDY ENROLLMENT: Enrollment in the study is expected to take approximately 6-9 months. Follow up will continue through 12 months, therefore, the duration of the study is approximately 18-21 months.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form;
2. Participant is 18 years of age and older;
3. Neurologically stable;
4. Ambulatory;
5. Symptomatic chronic venous insuSciency (CVI), with edema or pain, (CEAP classification of C3 or greater);
6. Flow-limiting venous outflow obstruction (>50%) within the intended target sites, defined by (a) a common femoral vein continuous waveform without respiratory variation on duplex ultrasound, or, (b) complete occlusion of any part of the iliofemoral tract as diagnosed on baseline duplex or axial imaging per local protocol; and
7. Target treatment IVC/Common Iliac confluence to the deep veins above the knee.

Exclusion Criteria:

1. Comorbidity risks which may limit longevity (<2 years life expectancy), would preclude open surgery, or would significantly increase risk for venous thrombo-embolism (VTE);
2. Invasive abdominal, pelvic or peripheral vascular surgery within 90 days of the procedure;
3. History of stroke within the last 6 months;
4. Known hypercoagulable states that, in the opinion of the Investigator, cannot be medically managed throughout the study period (i.e., known thrombophilia) including Heparin-induced thrombocytopenia (HIT) and antiphospholipid syndrome (APS);
5. Interventional procedure in the deep venous system (including stent placement) in the target limb or outflow vessels within 6 weeks of consent;
6. Acute deep venous thrombosis (DVT) in the index limb (not previously observed in the thrombus bearing segment) within 3 months of consent;
7. Inadequate inflow in the opinion of the investigator, that cannot be improved to the target vessel;
8. Flow-limiting venous outflow obstruction central to the target/treatment vessel that cannot be treated;
9. Pregnant and/or breastfeeding;
10. Patients with cognitive impairments who are unable to be consented;
11. Patient is enrolled in another clinical study that, in the opinion of the Investigator, may conflict with this study or compromise study results;
12. COPD or similar conditions (lung cancer, pulmonary hypertension, prior major lung surgery, emphysema, O2 dependency) that may, in the opinion of the investigator result in higher pulmonary risk; and
13. Patients considered to belong to a vulnerable population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-18 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint - Rates of all Adverse Events through 30-days post-index procedure | 30-days post-procedure
  The primary safety objective is procedural events defined as the rates of all adverse events occurring up to 30 days post-index procedure
Primary Efficacy Endpoint - Percent Lumen Gain in the Treated Vessel measured at time of procedure | Perioperative/Periprocedural
  The primary efficacy assessment includes the percent (%) lumen gain during the index procedure, which is measured using intravascular ultrasound (IVUS) at the time of the procedure

OTHER OUTCOMES:
Assessment of patency (using DUS) in the treated vessel | 30-days post-procedure
  Assessment of the treated venous segment patency (as defined by absence of occlusion and CD-TLR [clinically-driven target lesion revascularization]) at 30 days by DUS compared to baseline
Assessment of primary patency (defined as absence of occlusion and CD-TLR [clinically-driven target lesion revascularization]) in the vessel segment at all timepoints | 30-days, 90-days, 180-days and 365-days post-procedure
  Assessment of primary patency (as defined by absence of occlusion and CD-TLR) of the stented vessel segment via DUS comparison at post procedure and all follow ups 30-days, 90-days, 180-days and 365-days post-procedure
Assessment of secondary patency (defined as absence of occlusion and CD-TLR [clinically-driven target lesion revascularization]) in the stented vessel segment at all timepoints | 30-days, 90-days, 180-days and 365-days post-procedure
  Assessment of secondary patency (as defined by absence of occlusion and CD-TLR) of the stented segment via DUS at all follow-ups 30-days, 90-days, 180-days and 365-days post-procedure
Assessment of changes in Villalta Score at all timepoints | Baseline, 30-days, 90-days, 180-days and 365-days post-procedure
  Assessment of changes in the Villalta Score (Baseline through 365 days post-procedure); the score is a composite based on a rating score of absent (0), mild (1), moderate (2) and severe (3) for symptoms and clinical signs, and presence or absence of venous ulcers. A higher Villalta Score would indicate a worse outcome
Assessment of changes VCSS at all timepoints | Baseline, 30-days, 90-days, 180-days and 365-days post-procedure
  Assessment of changes in the VCSS Overall (Baseline through 365 days post-procedure); the score is a composite based on a rating score of none (0), mild (1), moderate (2) and severe (3) for symptoms and clinical signs, the number of active ulcers (0, 1, 2, >/=3), duration of ulcers (<3 months, >3 months but <1 year, not healed for >1 year), active ulcer size (diameter <2cm, diameter 2-6cm, and diameter >6cm), and use of compression therapy (not used (0), intermittent use of stockings (1), wears stockings most days (2), and full compliance (3)). A higher VCSS would indicate a worse outcome.
Assessment of VEINES QOL/Sym Score at all timepoints | Baseline, 30-days, 90-days, 180-days and 365-days post-procedure
  Assessment of changes in the VEINES QOL/Sym Score (Baseline through 365 days post-procedure); subjects are asked to complete a quality of life questionnaire consisting of 8 questions (26 items total). Each question consists of multiple response options for each category within the individual question. Of the 26 items in the questionnaire, 25 items are combined to create a summary score (VEINES-QOL). One item which asks about the time of day the leg problem is most intense provides only descriptive information and is not scored. A subset of ten of these items is used to create a symptom score (VEINES-Sym). For both the VEINES- QOL and VEINES-Sym scores, high values indicate better outcomes.
Rates of all Adverse Events through 365-days post-procedure | 365-days post-procedure]
  Rates of all adverse events occurring up to 365-days post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Black, MD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- St. Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No